CLINICAL TRIAL: NCT01472783
Title: Veliparib (ABT888) Monotherapy for Patients With BRCA Germline Mutation and Platinum-Resistant or Partially Platinum-Sensitive Relapse of Epithelial Ovarian Cancer
Brief Title: Veliparib Monotherapy for Relapsed Ovarian Cancer With BRCA Mutation
Acronym: Veli-BRCA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Veli-BRCA
Record Dates: First submitted 2011-11-02; First posted 2011-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Recurrent, Epithelial Ovarian Cancer
Keywords: BRCA1 mutation; BRCA2 mutation; Ovarian cancer; PARP inhibitor
MeSH Terms: conditions — Recurrence; Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Veliparib (Experimental)
  Interventions: Drug: Veliparib

INTERVENTIONS:
Drug: Veliparib — Veliparib (tablet) 300 mg twice daily on days 1-28 of 28 days cycles until progression, unacceptable toxicity or patient refusal.

SUMMARY:
The main purpose of this study is to investigate the effect of veliparib in ovarian cancer patients with known BRCA 1/2 mutations who do no longer respond to conventional chemotherapy.

DETAILED DESCRIPTION:
The side effects are modest, since PARP inhibitors affect cancer cells to a much larger extent than normal cells. The effect of this PARP-inhibiting treatment is evident although the greatest effect is seen in patients with mutations in BRCA genes. The reason for this is that BRCA deficient cancer cells are unable to repair both DNA double strand and single strand breaks and undergo apoptosis to a large extent.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed epithelial, primary fallopian or primary peritoneal cancer. Stages I-IV.
2. Patients with known germline BRCA1/2 mutations
3. Verified progression by either RECIST criteria and/or GCIG CA125 criteria after previous first line chemotherapy or progression after later lines of cytotoxic treatment.
4. Platinum resistance or partially platinum sensitive disease (Relapsed within six months of prior first line/later lines of platinum-based therapy or relapsed within six to twelve months of prior first line/later lines of platinum-based therapy)
5. Age ≥ 18 years.
6. Performance status 0-2.
7. Measurable disease by RECIST 1.1 or evaluable by CA125 GCIG criteria
8. Adequate bone marrow function, liver function, renal function and coagulation parameters (within 7 days prior to randomization):

   WBC ≥ 3.0 x 10^9/l or neutrophils (ANC) ≥ 1.5 x 10^9/l Platelet count ≥ 100 x 10^9/l Hemoglobin ≥ 9.7 g/dl (6 mmol/L) Serum bilirubin ≤ 1.5 x ULN Serum transaminases ≤ 2.5 x ULN Serum creatinine ≤ 1.5 x ULN
9. Written informed consent.
10. Tissue available for BRCAness analysis.

Exclusion Criteria:

1. Previous treatment with a PARP inhibitor.
2. Platinum-refractory disease (disease that progressed or was stable during prior platinum therapy)
3. Patients who have received (or are planning to receive) treatment with any other investigational regimen, or who have participated in another clinical trial within 28 days prior to entering this trial.
4. Pregnant or breast-feeding patients. For fertile women a negative pregnancy test at screening is mandatory.
5. Fertile patients not willing to use acceptable and safe methods of contraception during and for 6 months after treatment
6. Other present or previous malignancy except curatively treated cervical cancer stage I, non-melanotic skin cancer or other cancer with minimal risk of relapse.

   Curatively treated prior breast cancer is allowed if no relapse is suspected at time of inclusion.
7. CNS metastasis.
8. History of any chronic medical or psychiatric condition or laboratory abnormality that is not medically controlled or in the opinion of the Investigator may increase the risks associated with study drug administration. (e.g. diabetes, cardiac diseases, hypertension, renal or liver disease).
9. Allergy to the ingredients of the study medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose, dose limiting toxicity, recommended phase II dose. | 6 months
Phase II: Response rate | Every 3 months

SECONDARY OUTCOMES:
Progression free survival | Every 3 months
Overall survival | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Vejle Hospital, Vejle, Denmark
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark